CLINICAL TRIAL: NCT02672852
Title: BI 655066 / ABBV-066 (Risankizumab) Versus Placebo In a Multicenter Randomized Double-blind Study in Patients With Moderate to Severe Chronic Plaque Psoriasis Evaluating the Efficacy and Safety With Randomized Withdrawal and Re-treatment (IMMhance)
Brief Title: BI 655066 / ABBV-066 (Risankizumab) in Moderate to Severe Plaque Psoriasis With Randomized Withdrawal and Re-treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-992; 2014-005102-38 (EudraCT Number); 1311.4 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-05

CONDITIONS: Psoriasis
Keywords: ABBV-066; BI 655066; risankizumab
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risankizumab (Experimental): Participants randomized at Baseline to receive double-blind (DB) risankizumab 150 mg by subcutaneous injection at Weeks 0 and 4 (Part A1).
  Interventions: Drug: Risankizumab
- Placebo (Placebo Comparator): Participants randomized at Baseline to receive double-blind (DB) placebo by subcutaneous injection at Weeks 0 and 4 (Part A1).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risankizumab — Risankizumab administered by subcutaneous injection
  Other Names: BI 655066; ABBV-066; SKYRIZI
  Arms: Risankizumab
Drug: Placebo — Placebo for risankizumab administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
This was a multinational, multicenter, randomized, double-blind, placebo controlled study with randomized withdrawal and retreatment, evaluating the safety and efficacy of risankizumab 150 mg subcutaneous (SC) in participants with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
In Part A1, eligible participants were randomized at Baseline at a ratio of 4:1, stratified by weight and prior exposure to tumor necrosis factor antagonists to receive double-blind (DB) risankizumab 150 mg or placebo at Weeks 0 and 4. In Part A2, participants randomized at Baseline to receive DB placebo then received risankizumab 150 mg at Weeks 16 (Part A2) and at Week 28 and every 12 weeks up to 88 weeks (Part B); participants randomized to risankizumab 150 mg continued to receive risankizumab 150 mg at Week 16. Participants who received risankizumab in Part A and were nonresponders (sPGA >2) at Week 28 received risankizumab 150 mg at Week 28 and every 12 weeks up to 88 weeks (Part B). In Part B, participants who received risankizumab in Part A and were responders (sPGA ≤2) at Week 28, were rerandomized at a ratio of 1:2 to receive DB risankizumab 150 mg or placebo at Week 28 and every 12 weeks up to 88 weeks (Part B). Starting at Week 32, rerandomized participants who reached relapse (defined as sPGA ≥3) were switched to risankizumab 150 mg every 12 weeks.

ELIGIBILITY:
Inclusion criteria:

* Male or female participants. Woman of childbearing potential must be ready and willing to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1 percent per year when used consistently and correctly.
* Age ≥18 years at screening
* Have a diagnosis of chronic plaque psoriasis (with or without psoriatic arthritis) at least 6 months before the first administration of study drug. Duration of diagnosis may be reported by the participant.
* Have stable moderate to severe chronic plaque psoriasis with or without psoriatic arthritis at both Screening and Baseline (Randomization); Have an involved body surface area (BSA) ≥ 10% and Have a Psoriasis Area and Severity Index (PASI) ≥ 12 and Have a static Physician Global Assessment (sPGA) score of ≥ 3.
* Must be a candidate for systemic therapy or phototherapy for psoriasis treatment, as assessed by the investigator
* Signed and dated written informed consent prior to admission to the study and performance of any study procedures in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Participants with nonplaque forms of psoriasis (including guttate, erythrodermic, or pustular); current drug-induced psoriasis (including a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium); active ongoing inflammatory diseases other than psoriasis and psoriatic arthritis that might confound trial evaluations according to the investigators judgment.
* Previous exposure to ABBV-066
* Currently enrolled in another investigational study or less than 30 days (from screening) since completing another investigational study
* Use of any restricted medication as noted or any drug considered likely to interfere with the safe conduct of the study.
* Major surgery performed within 12 weeks prior to randomization or planned within 12 months after screening (e.g., hip replacement, removal aneurysm, stomach ligation).
* Known chronic or relevant acute infections such as active tuberculosis, human immunodeficiency virus (HIV), or viral hepatitis
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix
* Evidence of a current or previous disease (including chronic alcohol or drug abuse), medical condition other than psoriasis, surgical procedure (i.e., organ transplant), medical examination finding (including vital signs and electrocardiogram [ECG]), or laboratory value at the screening visit outside the reference range that in the opinion of the Investigator, is clinically significant and would make the study participant unable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data.
* History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Previous enrolment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Lebwohl MG, Soliman AM, Yang H, Wang J, Hagan K, Padilla B, Pinter A. Impact of Risankizumab on PASI90 and DLQI0/1 Duration in Moderate-to-Severe Psoriasis: A Post Hoc Analysis of Four Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2022 Feb;12(2):407-418. doi: 10.1007/s13555-021-00660-3. Epub 2021 Dec 18. PMID 34921669
- [Derived] Blauvelt A, Leonardi CL, Gooderham M, Papp KA, Philipp S, Wu JJ, Igarashi A, Flack M, Geng Z, Wu T, Camez A, Williams D, Langley RG. Efficacy and Safety of Continuous Risankizumab Therapy vs Treatment Withdrawal in Patients With Moderate to Severe Plaque Psoriasis: A Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2020 Jun 1;156(6):649-658. doi: 10.1001/jamadermatol.2020.0723. PMID 32267471
- [Derived] Suleiman AA, Khatri A, Oberoi RK, Othman AA. Exposure-Response Relationships for the Efficacy and Safety of Risankizumab in Japanese Subjects with Psoriasis. Clin Pharmacokinet. 2020 May;59(5):575-589. doi: 10.1007/s40262-019-00829-2. PMID 31667790
- [Derived] Suleiman AA, Minocha M, Khatri A, Pang Y, Othman AA. Population Pharmacokinetics of Risankizumab in Healthy Volunteers and Subjects with Moderate to Severe Plaque Psoriasis: Integrated Analyses of Phase I-III Clinical Trials. Clin Pharmacokinet. 2019 Oct;58(10):1309-1321. doi: 10.1007/s40262-019-00759-z. PMID 31054118
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A1: double-blind (DB) risankizumab or placebo (Weeks 0,4). Part A2 (Week 16) DB placebo to DB risankizumab; risankizumab continued risankizumab. Part B (Week 28) risankizumab responders rerandomized to DB risankizumab/placebo; risankizumab nonresponders continued risankizumab. Week 32: rerandomized relapsed switch risankizumab.
Groups:
- Placebo (Part A1): Participants randomized at Baseline to receive double-blind (DB) placebo at Weeks 0 and 4 (Part A1).
- Risankizumab (Part A1): Participants randomized at Baseline to receive double-blind (DB) risankizumab 150 mg at Weeks 0 and 4 (Part A1).
- Placebo/Risankizumab Part A2/Part B: Participants randomized at Baseline to receive double-blind (DB) placebo then received DB risankizumab 150 mg at Weeks 16 (Part A2) and at Week 28 and every 12 weeks up to 88 weeks (Part B).
- Risankizumab/Risankizumab Part A2: Participants randomized at Baseline to receive double-blind (DB) risankizumab then received DB risankizumab 150 mg at Weeks 16 (Part A2).
- Risankizumab/Placebo (Part B; Rerandomized Responders): Participants who received risankizumab in Part A and were responders (sPGA 0 or 1) at Week 28, and rerandomized to receive placebo at Week 28 and every 12 weeks up to Week 88 (Part B).
- Risankizumab/Risankizumab (Part B; Rerandomized Responders): Participants who received risankizumab in Part A and were responders (sPGA 0 or 1) at Week 28, and rerandomized to receive risankizumab 150 mg at Week 28 and every 12 weeks up to Week 88 (Part B).
- Risankizumab/Risankizumab Part B (Nonresponders): Participants who received risankizumab in Part A and were nonresponders (sPGA ≥2) at Week 28 received risankizumab 150 mg at Week 28 and every 12 weeks up to 88 weeks (Part B).
Period: Part A1
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1) | Placebo/Risankizumab Part A2/Part B | Risankizumab/Risankizumab Part A2 | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders) | Risankizumab/Risankizumab Part B (Nonresponders)
Started | 100 | 407 | 0 | 0 | 0 | 0 | 0
Completed | 97 | 403 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Worsening | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part A2
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1) | Placebo/Risankizumab Part A2/Part B | Risankizumab/Risankizumab Part A2 | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders) | Risankizumab/Risankizumab Part B (Nonresponders)
Started | 0 (Participants that completed Part A1 continued on to Part A2.) | 0 (Participants that completed Part A1 continued on to Part A2.) | 93 (Participants that completed Part A1 continued on to Part A2.) | 403 (Participants that completed Part A1 continued on to Part A2.) | 0 | 0 | 0
Completed | 0 | 0 | 83 | 399 | 0 | 0 | 0
Not Completed | 0 | 0 | 10 | 4 | 0 | 0 | 0
Not completed — Disease worsening | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Not entered in Part B | 0 | 0 | 0 | 4 | 0 | 0 | 0
Period: Part B
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1) | Placebo/Risankizumab Part A2/Part B | Risankizumab/Risankizumab Part A2 | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders) | Risankizumab/Risankizumab Part B (Nonresponders)
Started | 0 | 0 | 0 (Participants that completed Part A2 continued on to Part B.) | 0 (Participants that completed Part A2 continued on to Part B.) | 225 (Participants that completed Part A2 continued on to Part B.) | 111 (Participants that completed Part A2 continued on to Part B.) | 63 (Participants that completed Part A2 continued on to Part B.)
Completed | 0 | 0 | 0 | 0 | 209 | 100 | 51
Not Completed | 0 | 0 | 0 | 0 | 16 | 11 | 12
Not completed — Disease worsening | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Worsening pre-existing condition | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other adverse event | 0 | 0 | 0 | 0 | 3 | 5 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5 | 0 | 7
Not completed — Other | 0 | 0 | 0 | 0 | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population in Part A1 (ITT_A1): All participants who were randomized at Baseline
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1) | Total
Number analyzed (Participants) | 100 | 407 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (13.78) | 49.6 (13.17) | 49.2 (13.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 124 | 151
  Male | 73 | 283 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 45 | 56
  Not Hispanic or Latino | 89 | 362 | 451
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 64 | 79
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 2 | 18 | 20
  White | 82 | 320 | 402
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 90% Improvement Psoriasis Area and Severity Index (PASI) Score (PASI90) From Baseline to Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Non-responder imputation (NRI) was used for missing data.
Time Frame: Baseline, Week 16
Population: Intent to treat (ITT) Population in Part A1(ITT_A1): all participants who were randomized at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1)
Number analyzed (Participants) | 100 | 407
percentage of participants | 2.0 | 73.2
Statistical Analysis 1: Comparison: Placebo (Part A1) vs Risankizumab (Part A1); Across strata, P value was calculated from the Cochran-Mantel-Haenszel (CMH) test adjusted for strata. Within each stratum, P value was calculated based on the chi-square test (or Fisher's exact test if ≥25% of the cells had expected cell count <5); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 70.8, 95% CI 2-sided [65.7 to 76.0]

2. Primary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) Score of Clear or Almost Clear at Week 16
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5. NRI was used for missing data.
Time Frame: Week 16
Population: ITT Population in Part A1(ITT_A1)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1)
Number analyzed (Participants) | 100 | 407
percentage of participants | 7.0 | 83.5
Statistical Analysis 1: Comparison: Placebo (Part A1) vs Risankizumab (Part A1); Across strata, P value was calculated from the CMH test adjusted for strata. Within each stratum, P value was calculated based on the chi-square test (or Fisher's exact test if ≥25% of the cells had expected cell count <5); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 76.5, 95% CI 2-sided [70.4 to 82.5]

3. Primary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 52
Description: as for outcome 2
Time Frame: Week 52
Population: ITT Population in Part B for re-randomized participants (ITT_B_R): All participants who were randomized to Arm 1 at Baseline and re randomized at Week 28.
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders)
Number analyzed (Participants) | 225 | 111
percentage of participants | 61.3 | 87.4
Statistical Analysis 1: Comparison: Risankizumab/Placebo (Part B; Rerandomized Responders) vs Risankizumab/Risankizumab (Part B; Rerandomized Responders); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 25.9, 95% CI 2-sided [17.3 to 34.6]

4. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Population: ITT Population in Part A1 (ITT_A1)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1)
Number analyzed (Participants) | 100 | 407
percentage of participants | 8.0 | 88.7
Statistical Analysis 1: Comparison: Placebo (Part A1) vs Risankizumab (Part A1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 80.6, 95% CI 2-sided [74.5 to 86.6]

5. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI Score (PASI100) at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Population: ITT Population in Part A1 (ITT_A1)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1)
Number analyzed (Participants) | 100 | 407
percentage of participants | 1.0 | 47.2
Statistical Analysis 1: Comparison: Placebo (Part A1) vs Risankizumab (Part A1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 45.5, 95% CI 2-sided [40.3 to 50.8]

6. Secondary Outcome: Percentage of Participants Achieving an sPGA Score of Clear at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: ITT Population in Part A1 (ITT_A1)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1)
Number analyzed (Participants) | 100 | 407
percentage of participants | 1.0 | 46.4
Statistical Analysis 1: Comparison: Placebo (Part A1) vs Risankizumab (Part A1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 44.8, 95% CI 2-sided [39.5 to 50.0]

7. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16
Description: The DLQI is a 10-question questionnaire that asks the participant to evaluate the degree that psoriasis has affected their quality of life in the last week and includes 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). Responses to each domain are not relevant (0), not at all (0), a little (1), a lot (2), and very much (3). The DLQI is calculated by summing the scores of the questions and ranges from 1 to 30, where 0-1 = no effect on patient's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on patient's life. The higher the score, the more the quality of life is impaired. NRI was used for missing data.
Time Frame: Week 16
Population: ITT Population in Part A1 (ITT_A1)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1)
Number analyzed (Participants) | 100 | 407
percentage of participants | 3.0 | 65.4
Statistical Analysis 1: Comparison: Placebo (Part A1) vs Risankizumab (Part A1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 62.1, 95% CI 2-sided [56.4 to 67.9]

8. Secondary Outcome: Percentage of Participants Achieving an sPGA Score of Clear or Almost Clear at Week 104
Description: as for outcome 2
Time Frame: Week 104
Population: ITT Population in Part B for re-randomized participants (ITT_B_R)
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders)
Number analyzed (Participants) | 225 | 111
percentage of participants | 7.1 | 81.1
Statistical Analysis 1: Comparison: Risankizumab/Placebo (Part B; Rerandomized Responders) vs Risankizumab/Risankizumab (Part B; Rerandomized Responders); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 73.9, 95% CI 2-sided [66.0 to 81.9]

9. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 52
Description: as for outcome 4
Time Frame: Week 52
Population: ITT Population in Part B for re-randomized participants (ITT_B_R)
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders)
Number analyzed (Participants) | 225 | 111
percentage of participants | 71.6 | 92.8
Statistical Analysis 1: Comparison: Risankizumab/Placebo (Part B; Rerandomized Responders) vs Risankizumab/Risankizumab (Part B; Rerandomized Responders); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 21.2, 95% CI 2-sided [13.7 to 28.7]

10. Secondary Outcome: Percentage of Participants Achieving 90% Improvement in PASI Score (PASI90) at Week 52
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 52
Population: ITT Population in Part B for re-randomized participants (ITT_B_R)
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders)
Number analyzed (Participants) | 225 | 111
percentage of participants | 52.4 | 85.6
Statistical Analysis 1: Comparison: Risankizumab/Placebo (Part B; Rerandomized Responders) vs Risankizumab/Risankizumab (Part B; Rerandomized Responders); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 33.1, 95% CI 2-sided [24.0 to 42.2]

11. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI Score (PASI100) at Week 52
Description: as for outcome 5
Time Frame: Week 52
Population: ITT Population in Part B for re-randomized participants (ITT_B_R)
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders)
Number analyzed (Participants) | 225 | 111
percentage of participants | 30.2 | 64.0
Statistical Analysis 1: Comparison: Risankizumab/Placebo (Part B; Rerandomized Responders) vs Risankizumab/Risankizumab (Part B; Rerandomized Responders); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted percentage difference = 33.7, 95% CI 2-sided [23.2 to 44.2]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 15 weeks after the last dose of study drug (up to 103 weeks).
Description: TEAEs and TESAEs: defined as any adverse event (AE) or serious adverse event (SAE) with onset or worsening reported by participant from time to first dose of study drug administered within 15 weeks following discontinuation of risankizumab administration or, for AEs presented by study Part, from first dose in the study Part until prior to first dose in the subsequent study Part (Part A1=from Week 0 until prior to Week 16 dose; Part B=from Week 28 to 15 weeks after last dose at [up to Week 103]).
Groups:
- Placebo (Part A1): All participants randomized at Baseline to receive double-blind (DB) placebo at Weeks 0 and 4 (Part A1).
- Risankizumab (Part A1): All participants randomized at Baseline to receive double-blind (DB) risankizumab 150 mg at Weeks 0 and 4 (Part A1).
- Any Risankizumab: Participants who received at least one dose of risankizumab during the study.
Arm/Group | Placebo (Part A1) | Risankizumab (Part A1) | Risankizumab/Placebo (Part B; Rerandomized Responders) | Risankizumab/Risankizumab (Part B; Rerandomized Responders) | Any Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/407 | 0/225 | 2/111 | 4/500
Serious Adverse Events (participants affected / at risk) | 8/100 | 8/407 | 17/225 | 13/111 | 55/500
Other Adverse Events (participants affected / at risk) | 17/100 | 52/407 | 92/225 | 52/111 | 242/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A1) (N=100) | Risankizumab (Part A1) (N=407) | Risankizumab/Placebo (Part B; Rerandomized Responders) (N=225) | Risankizumab/Risankizumab (Part B; Rerandomized Responders) (N=111) | Any Risankizumab (N=500)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Benign familial pemphigus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Huntington's disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol detoxification (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A1) (N=100) | Risankizumab (Part A1) (N=407) | Risankizumab/Placebo (Part B; Rerandomized Responders) (N=225) | Risankizumab/Risankizumab (Part B; Rerandomized Responders) (N=111) | Any Risankizumab (N=500)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 8 (10) | 7 (8) | 22 (24)
Nasopharyngitis (Infections and infestations) | 6 (6) | 21 (21) | 45 (53) | 23 (36) | 116 (170)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 6 (6) | 23 (29) | 16 (19) | 77 (97)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 13 (16) | 10 (10) | 35 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 12 (13) | 4 (7) | 28 (31)
Headache (Nervous system disorders) | 0 (0) | 14 (15) | 7 (9) | 8 (15) | 34 (47)
Psoriasis (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 8 (8) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-10-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT02672852/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT02672852/SAP_001.pdf